CLINICAL TRIAL: NCT05950516
Title: Efficacy and Safety of Semaglutide Injection (QLG2065) vs. Ozempic® as add-on to Metformin in Type 2 Diabetics.
Brief Title: Efficacy and Safety of Semaglutide Ingection in Subjects With Type 2 Diabetes
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QLG2065-301
Record Dates: First submitted 2023-07-11; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QLG2065 (Experimental): Up to 1.0 mg semaglutide (QLG2065)
  Metformin ≥ 1500 mg/day (or maximum tolerated dose ≥ 1000 mg/day).
  Interventions: Drug: Semaglutide
- Ozempic (Active Comparator): Up to 1.0 mg semaglutide (Ozempic)
  Metformin ≥ 1500 mg/day (or maximum tolerated dose ≥ 1000 mg/day).
  Interventions: Drug: Semaglutide Pen Injector [Ozempic]

INTERVENTIONS:
Drug: Semaglutide — Up to 1.0 mg semaglutide injected subcutaneously once-weekly for 32 weeks
  Other Names: QLG2065
  Arms: QLG2065
Drug: Semaglutide Pen Injector [Ozempic] — Up to 1.0 mg semaglutide injected subcutaneously once-weekly for 32 weeks
  Other Names: Ozempic Injectable Product
  Arms: Ozempic

SUMMARY:
To evaluate the similarity of the efficacy and safety of semaglutide injection (QLG2065) vs. Ozempic® in patients with type 2 diabetes mellitus (T2DM) with poor blood glucose control after metformin treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age ≥ 18 years and ≤75 years old at the time of screening.
2. Subjects diagnosed with type 2 diabetes for at least 6 months (WHO, 1999)
3. Within 60 days before screening, subjects received stable treatment with only metformin ≥ 1500 mg/day (or maximum tolerated dose ≥ 1000 mg/day), or receive combination metformin (dose ≥ 750 mg/day) and another OAD (alpha-glucosidase inhibitors, sulfonylureas, glinides, SGLT-2i or thiazolidinedione), stable treatment is defined as unchanged medication and daily doses;
4. At the time of screening, for those who have previously been treated with metformin alone, HbA1c ≥ 7.0% and ≤ 11.0%（local lab）; for those who have previously used metformin in combination with another OAD treatment, HbA1c ≥ 7.0% and ≤10.0%（local lab）;
5. BMI≥18.5kg/m2 and ≤35 kg/m2
6. Subjects voluntarily participate in this research, can communicate well with researchers, are willing to maintain the same diet and exercise habits throughout the study, and sign an informed consent form (ICF) .
7. At baseline，HbAlc ≥ 7.0% and ≤ 11.0%（cental lab）

Exclusion Criteria:

1. Known or suspected hypersensitivity to any GLP-1RA or related products, or allergic constitution
2. Treatment with GLP-1RA, DPP-4 inhibitor, or insulin in a period of 60 days before screening. An exception is short-term insulin therapy (≤7 days in total).
3. History of chronic or acute pancreatitis
4. Screening calcitonin value ≥ 50 ng/L (pg/mL)
5. Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN 2)
6. Have a history of major cardiovascular and cerebrovascular diseases within 90 days before screening.
7. Known proliferative retinopathy or maculopathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Estimated)
Dates: Start 2023-07-10 (Estimated); Primary Completion 2024-11-24 (Estimated); Study Completion 2025-01-22 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | Week 33
  Change from baseline (week 1) to week 33 in glycosylated haemoglobin (HbA1c) was evaluated

SECONDARY OUTCOMES:
Change in HbA1c | Week 21
  Change from baseline (week 1) to week 21 in glycosylated haemoglobin (HbA1c) was evaluated
Percentage of Participants Who Achieved HbA1c <7.0% , HbA1c ≤6.5% | Week 21, 33
  Percentage of participants who achieved HbA1c < 7.0%, HbA1c ≤6.5% is presented
Change in Fasting Glucose | Week 21, 33
  Change from baseline (week 1) to week 21, 33 in Fasting Glucose was evaluated
Change in Body Weight | Week 21, 33
  Change from baseline (week 1) to week 21, 33 in body weight was evaluated
Percentage of Participants That Achieved Body Weight Loss ≥5% | Week 21, 33
  Percentage of participants losing ≥5% of baseline body weight is presented

CONTACTS AND LOCATIONS:
Overall Officials: Jiajun Zhao, Principal Investigator — Shandong Provincial Hospital
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No